CLINICAL TRIAL: NCT02210871
Title: A Multi-centre, Open-label, Parallel-group Trial Investigating the Pharmacokinetics, Safety and Tolerability After a Single Subcutaneous Injection of Semaglutide in Subjects With Mild, Moderate or Severe Hepatic Impairment Compared to Subjects With Normal Hepatic Function
Brief Title: Investigating the Pharmacokinetics, Safety and Tolerability After a Single Subcutaneous Injection of Semaglutide in Subjects With Mild, Moderate or Severe Hepatic Impairment Compared to Subjects With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9535-3651; U1111-1149-3924 (Other: WHO); 2009-011673-33 (EudraCT Number)
Record Dates: First submitted 2014-08-06; First posted 2014-08-07 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Hepatic Impaired
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Normal hepatic function (Experimental)
  Interventions: Drug: semaglutide
- Mild hepatic impairment (Experimental)
  Interventions: Drug: semaglutide
- Moderate hepatic impairment (Experimental)
  Interventions: Drug: semaglutide
- Severe hepatic impairment (Experimental)
  Interventions: Drug: semaglutide

INTERVENTIONS:
Drug: semaglutide — All subjects will be treated with a single subcutane (s.c., under the skin) injection of 0.5 mg semaglutide.

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the pharmacokinetics (the exposure of the trial drug in the body), safety and tolerability after a single injection of semaglutide in subjects with mild, moderate or severe hepatic impairment compared to subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age at least 18 years at the time of signing informed consent
* Body mass index (BMI) 18.5-40.0 kg/m^2 (both inclusive)
* Only for subjects with hepatic impairment (mild, moderate and severe): A diagnosis of cirrhosis due to parenchymal liver disease, classified as Child-Pugh grade A,B or C as assessed by investigator and which is confirmed and documented by medical history, physical examination and at least one of the following: hepatic ultrasound,computerised axial tomography (CT) scan, magnetic resonance imaging (MRI), and/or liver biopsy
* Only for subjects with normal hepatic function: Subjects who are judged to be in good general health based on physical examination, medical history, ECG, vital signs, and the results of biochemistry, coagulation, haematology tests and urinalysis performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential not using an adequate contraceptive method throughout the trial including the follow-up period (adequate contraceptive measures as required by local regulation or practice)
* Uncontrolled hypertension (defined as systolic blood pressure above or equal to 180 mmHg and/or diastolic blood pressure above or equal to 100 mmHg). If white-coat hypertension is suspected at the screening visit a repeated measurement at the screening visit is allowed
* Mental inability, unwillingness or language barrier precluding adequate understanding of or compliance with trial procedures
* Donation of any blood or plasma in the past month or in excess of 400 mL within the 3 months preceding screening, or surgery or trauma with more than 400 mL blood loss within the 3 months preceding screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-08-07 (Actual); Primary Completion 2015-06-03 (Actual); Study Completion 2015-06-03 (Actual)

PRIMARY OUTCOMES:
Area under the semaglutide plasma concentration-time curve | Day 1 - day 36

SECONDARY OUTCOMES:
Maximum observed semaglutide plasma concentration | Day 1 - day 36
Number of treatment emergent adverse events (TEAEs) | Day 1 - day 36

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry GCR, 1452, Study Director — Novo Nordisk A/S
Locations (3):
- Poland (2):
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wołomin
- Novo Nordisk Investigational Site, Bratislava, Slovakia

REFERENCES:
- [Result] Jensen L, Kupcova V, Arold G, Pettersson J, Hjerpsted JB. Pharmacokinetics and tolerability of semaglutide in people with hepatic impairment. Diabetes Obes Metab. 2018 Apr;20(4):998-1005. doi: 10.1111/dom.13186. Epub 2018 Jan 17. PMID 29205786
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com